CLINICAL TRIAL: NCT05805501
Title: A Randomized Open Label Phase II Study of Immune Checkpoint Inhibitor Combinations With Axitinib in Patients With Previously Untreated Locally Advanced Unresectable or Metastatic Renal Cell Carcinoma
Brief Title: A Study of Immune Checkpoint Inhibitor Combinations With Axitinib in Participants With Untreated Locally Advanced Unresectable or Metastatic Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO43936
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Tiragolumab; pembrolizumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Tobemstomig + Axitinib) (Experimental): Participants will receive intravenous (IV) tobemstomig every three weeks (Q3W) on Day 1 of each 21-day cycle. Participants will also receive oral (PO) axitinib twice daily (BID).
  Interventions: Drug: Tobemstomig; Drug: Axitinib
- Arm B (Tobemstomig + Tiragolumab + Axitinib) (Experimental): Participants will receive IV tobemstomig followed by IV tiragolumab Q3W on Day 1 of 21-day cycle. Participants will also receive axitinib PO BID.
  Interventions: Drug: Tobemstomig; Drug: Tiragolumab; Drug: Axitinib
- Control Arm (Pembrolizumab + Axitinib) (Active Comparator): Participants will receive IV pembrolizumab Q3W on Day 1 of each 21-day cycle. Participants will also receive axitinib PO BID.
  Interventions: Drug: Pembrolizumab; Drug: Axitinib

INTERVENTIONS:
Drug: Tobemstomig — Participants will receive IV tobemstomig Q3W.
  Other Names: RO7247669
  Arms: Arm A (Tobemstomig + Axitinib); Arm B (Tobemstomig + Tiragolumab + Axitinib)
Drug: Tiragolumab — Participants will receive IV tiragolumab Q3W.
  Arms: Arm B (Tobemstomig + Tiragolumab + Axitinib)
Drug: Pembrolizumab — Participants will receive IV pembrolizumab Q3W.
  Other Names: Keytruda
  Arms: Control Arm (Pembrolizumab + Axitinib)
Drug: Axitinib — Participants will receive axitinib PO BID.
  Other Names: Inlyta

SUMMARY:
This study will evaluate the safety of tobemstomig (RO7247669) in combination with axitinib alone or with tiragolumab (anti-TIGIT) and axitinib as compared to pembrolizumab and axitinib in participants with previously untreated, unresectable locally advanced or metastatic clear-cell renal cell carcinoma (ccRCC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* International Metastatic RCC Database Consortium (IMDC) risk intermediate (score of 1 or 2) or poor (score of 3-6)
* Measurable disease with at least one measurable lesion
* Histologically confirmed ccRCC with or without sarcomatoid features
* Negative for HIV, hepatitis B, or hepatitis C virus (HCV)

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within 90 days after the final dose of tiragolumab, 4 months after the final dose of tobemstomig (RO7249669) and pembrolizumab, or for 1 week after the final dose of axitinib, whichever occurs last
* Inability to swallow a tablet or malabsorption syndrome
* Prior treatment for localized and/or metastatic RCC with systemic RCC-directed therapy, including T-cell costimulating or immune checkpoint blockade therapies
* Ongoing use or anticipated need for treatment with a strong CYP3A4/5 inhibitor or inducer
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Uncontrolled or symptomatic hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Moderate to severe hepatic impairment (Child-Pugh B or C)
* Uncontrolled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant cardiovascular/cerebrovascular disease within 3 months (12 months for UK participants) prior to randomization
* History of clinically significant ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* History of congenital QT syndrome
* Resting heart rate (HR) > 100 bpm (or clinically significant tachycardia)
* Stroke (including transient ischemic attack), myocardial infarction, or other symptomatic ischemic event, or thromboembolic event (e.g., deep venous thrombosis [DVT], pulmonary embolism [PE]) within 3 months (12 months for UK participants) before randomization
* Significant vascular disease (e.g., aortic aneurysm or arterial dissection requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of Cycle 1
* Tumors invading pulmonary blood vessels, cavitating pulmonary lesions or known endobronchial disease
* Tumor invading the gastrointestinal (GI) tract, including abdominal or tracheoesophageal fistulas
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Active peptic ulcer disease, acute pancreatitis, acute obstruction of the pancreatic or biliary duct, appendicitis, cholangitis, cholecystitis, diverticulitis, gastric outlet obstruction
* Intra-abdominal abscess within 6 months before initiation of study treatment
* Clinical signs or symptoms of GI obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of bleeding diathesis or significant coagulopathy
* Grade ≥ 3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment
* Clinically significant hematuria, hematemesis, hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, coagulopathy, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 3 months before initiation of study treatment
* Active or history of autoimmune disease or immune deficiency
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* History of another primary malignancy other than RCC within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%)
* Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live, attenuated vaccine will be required during the study
* Active tuberculosis (TB)
* Severe infection within 4 weeks prior to initiation of study treatment
* Participants with active Epstein-Barr virus (EBV) infection or known or suspected chronic active EBV infection at screening
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Known hypersensitivity to Chinese hamster *ovary cell products or to any component of tobemstomig, tiragolumab, pembrolizumab, or axitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | Up to a maximum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (43):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Irvine Medical Center, Orange, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
- Sunshine Coast University Hospital, Birtinya, Queensland, Australia
- China (4):
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Tianjin Cancer Hospital, Tianjin
- France (6):
  - Institut Sainte Catherine, Avignon
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum "Carl Gustav Carus", Dresden
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar der TU München, München
  - Studienpraxis Urologie, Nürtingen
  - Universitätsklinikum Ulm, Ulm
- Poland (4):
  - Szpital Specjalistyczny Podkarpacki O?rodek Onkologiczny, Brzozów
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu, Późna
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - Barts & London School of Med, London
  - Christie Hospital Nhs Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing